CLINICAL TRIAL: NCT01074853
Title: Evaluation of Beta Blockers for the Treatment of Asthma. A Randomised Controlled Trial of Propranolol
Brief Title: Beta Blockers for the Treatment of Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Principal Investigator, Brian J Lipworth, Professor, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PAW004
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Experimental): Chronic dose escalation of propranolol over period of 6 to 8 weeks.
  Interventions: Drug: propranolol
- Placebo (Placebo Comparator): Matched placebo used for dose escalation period of 6 to 8 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: propranolol — 10mg twice daily escalated to 80mg once daily
  Arms: Propranolol
Drug: placebo — Matched placebo
  Arms: Placebo

SUMMARY:
Current asthma medicines include inhalers. A common inhaler used in asthma is called a beta-agonist (for example salbutamol). They improve asthma symptoms by stimulating areas in the human airway resulting in widening of the human airway. Although these drugs are useful after the first dose, longterm use can cause worsening asthma symptoms.

Beta-blockers are the complete opposite type of medication. Just now they are avoided in patients with asthma as after the first dose they can cause airway narrowing and cause an asthma attack.

New research has suggested that long term use of beta-blockers can reduce airway inflammation which can improve asthma control and improve symptoms.

This research was done in asthmatic patients who didn't need inhaled steroids to control their asthma. What the investigators want to do is see if the same benefit of beta-blocker use is asthma can be seen in people who take inhaled steroids.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers with stable mild intermittent or mild persistent asthma.
* Stable defined as: FEV1 (Forced Expiratory Volume in 1second) >80% predicted with diurnal FEV1 variation <30% when LABA (Long Acting Beta Agonist) washed out.
* Methacholine PC20 <4mg/ml.
* Ability to perform spirometry, IOS (Impulse Oscillometry), bronchial challenge and all domiciliary measurements.
* Ability to obtain Informed consent.
* Mild to Moderate Asthmatics taking ≤1000μg BDP (Beclomethasone Diproprionate) per day or equivalent.
* Withhold LABAs for 1 week prior to study.

Exclusion Criteria:

* Uncontrolled symptoms of asthma.
* Resting BP (Blood Pressure) <110 systolic or HR (Heart Rate)<60.
* Pregnancy or lactation.
* Known or suspected sensitivity to the IMP (Investigational Medicinal Product)(s).
* Inability to comply with protocol.
* Any degree of heart block.
* Rate limiting medication including β blockers, rate limiting Calcium - Channel Blockers and Amiodarone.
* Any other clinically significant medical condition that may either endanger the health or safety of the participant, or jeopardise the protocol.
* An asthma exacerbation within the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To establish effects of chronic dosing with 'beta-blockers' on airway tone and hyperreactivity in mild asthmatics. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Lipworth, MD, Principal Investigator — University of Dundee
Locations (1):
- Asthma and Allergy Research Group, Unviersity of Dundee, Dundee, United Kingdom

REFERENCES:
- [Result] Short PM, Williamson PA, Anderson WJ, Lipworth BJ. Randomized placebo-controlled trial to evaluate chronic dosing effects of propranolol in asthma. Am J Respir Crit Care Med. 2013 Jun 15;187(12):1308-14. doi: 10.1164/rccm.201212-2206OC. PMID 23593932
- [Derived] Short PM, Anderson WJ, Manoharan A, Lipworth BJ. Usefulness of impulse oscillometry for the assessment of airway hyperresponsiveness in mild-to-moderate adult asthma. Ann Allergy Asthma Immunol. 2015 Jul;115(1):17-20. doi: 10.1016/j.anai.2015.04.022. PMID 26123421